CLINICAL TRIAL: NCT01970345
Title: A Pilot Treatment Study of Insulin-Like Growth Factor-1 (IGF-1) in Autism Spectrum Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision made to terminate due to difficulty in procurement of adequate supply of treatment drug. Decision made on April 2023 to terminate study.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Autism Science Foundation (Other)
Responsible Party: Principal Investigator, Alexander Kolevzon, Clinical Director, Seaver Autism Center for Research and Treatment, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 13-1206
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; IGF-1
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Insulin-Like Growth Factor I; mecasermin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGF-1 (Experimental): Randomized, placebo-controlled, crossover format with 12 weeks in each treatment arm (IGF-1 and placebo), separated by a four-week wash-out phase.
  Dose titration will be initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Doses may be decreased according to tolerability by 0.04 mg/kg per dose. Medication will be administered twice daily with meals, and preprandial glucose monitoring will be performed by parents at treatment initiation, prior to each injection, and until a well tolerated dose is established.
  Interventions: Drug: IGF-1
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo/saline

INTERVENTIONS:
Drug: IGF-1 — IGF-1 is an FDA-approved (IND exemption #113450), commercially available compound that crosses the blood-brain barrier and has beneficial effects on synaptic development by promoting neuronal cell survival, synaptic maturation, and synaptic plasticity.
  Other Names: Increlex; mecasermin
  Arms: IGF-1
Drug: Placebo/saline — Placebo
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The proposed project will pilot the use of IGF-1 as a novel treatment for core symptoms of autism. We will use a double-blind, placebo-controlled crossover trial design in five children with autism to evaluate the impact of IGF-1 treatment on autism-specific impairments in socialization, language, and repetitive behaviors. We expect to provide evidence for the safety and feasibility of IGF-1 in ameliorating social withdrawal in children with Autistic Disorder. Further, we expect to demonstrate that IGF-1 is associated with improvement on secondary outcomes of social impairment, language delay, and repetitive behavior, as well as on functional outcomes of global severity.

DETAILED DESCRIPTION:
IGF-1 is an FDA approved, commercially available compound that crosses the blood-brain barrier and has beneficial effects on synaptic development by promoting neuronal cell survival, synaptic maturation, and synaptic plasticity. IGF-1 is effective in reversing mouse and neuronal models of Rett syndrome and Phelan McDermid syndrome, both single gene causes of ASD and may therefore be effective in treating autism spectrum disorders (ASD) more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for Autism Spectrum Disorder confirmed by the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule- Generic (ADOS-G)
* Children between the ages of 5-12 years of age
* Language delay (lack of fluent phrase speech) reflected by use of ADOS Module 1 or 2
* Must be on stable medication regimens for at least three months prior to enrollment, assuming the concomitant medication is safe for use with IGF-1

Exclusion Criteria:

* Closed epiphyses
* Active or suspected neoplasia
* Intracranial hypertension
* Hepatic insufficiency
* Renal insufficiency
* Cardiomegaly/valvulopathy
* History of allergy to IGF-1
* Patients with comorbid conditions deemed too medically compromised to tolerate the risk of experimental treatment with IGF-1

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Long J, Liao X, Han K, Niu M, Chen J, Wang X, Liu J, Zhang Y, Zhang H. Association of Thyroid Hormone and Insulin-Like Growth Factor-1 Levels With Autism Spectrum Disorders: A Systematic Review and Meta-Analysis. Autism Res. 2025 Jul;18(7):1497-1512. doi: 10.1002/aur.70052. Epub 2025 May 12. PMID 40351246
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Decision made to terminate due to difficulty in procurement of adequate supply of treatment drug. Decision made on April 2023 to terminate study. However last participant visit was Sept 2017.
Groups:
- IGF-1 Then Placebo; Placebo Then IGF-1: Randomized, placebo-controlled, crossover format with 12 weeks in each treatment arm (IGF-1 and placebo), separated by a four-week wash-out phase.
  IGF-1: Dose titration initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Doses may be decreased according to tolerability by 0.04 mg/kg per dose. Medication will be administered twice daily with meals, and pre-prandial glucose monitoring will be performed by parents at treatment initiation, prior to each injection, and until a well-tolerated dose is established.
  Placebo: Matching Placebo
Period: First Treatment Phase 12 Weeks
Arm/Group | IGF-1 Then Placebo | Placebo Then IGF-1
Started | 1 | 2
Completed | 0 | 1
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Crossover Washout Period 4 Weeks
Arm/Group | IGF-1 Then Placebo | Placebo Then IGF-1
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: Second Treatment Phase 12 Weeks
Arm/Group | IGF-1 Then Placebo | Placebo Then IGF-1
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Children With Autism Spectrum Disorders: Randomized, placebo-controlled, crossover format with 12 weeks in each treatment arm (IGF-1 and placebo), separated by a four-week wash-out phase.
Arm/Group | Children With Autism Spectrum Disorders
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist - Social Withdrawal Subscale
Description: Aberrant Behavior Checklist - Social Withdrawal Subscale has16 items, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Total Subscale scores range from 0 to 48. Higher score indicates poorer health outcomes.
Time Frame: Phase 1 - Week 4 and 12, Phase 2 - Week 4 and 8
Population: Results for participants who were still on study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IGF-1: IGF-1: Dose titration initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Doses may be decreased according to tolerability by 0.04 mg/kg per dose. Medication will be administered twice daily with meals, and pre-prandial glucose monitoring will be performed by parents at treatment initiation, prior to each injection, and until a well-tolerated dose is established.
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale
  Week 4, phase 1 | 20 (NA) — N=1 therefore there is no measure of dispersion | 20 (18.4)
  Week 12, Phase 1: number analyzed (Participants) | 0 | 1
  Week 12, Phase 1 |  | 4 (NA) — N=1 therefore there is no measure of dispersion
  Week 4, phase 2: number analyzed (Participants) | 1 | 0
  Week 4, phase 2 | 3 (NA) — N=1 therefore there is no measure of dispersion |
  Week 8, Phase 2: number analyzed (Participants) | 1 | 0
  Week 8, Phase 2 | 2 (NA) — N=1 therefore there is no measure of dispersion |

2. Secondary Outcome: Social Pervasive Developmental Disorder-Behavior Inventory (PDDBI)
Description: Social Pervasive Developmental Disorder-Behavior Inventory (PDDBI) - Each item is marked as "0" (does not show the behavior), "1" (rarely shows the behavior), "2" (sometimes/partially shows the behavior), "3" (usually/typically shows the behavior), or "?" (uncertain/don't understand).
  The Sensory, Ritual, Social Pragmatic, Semantic Pragmatic, Arouse, Specific Fears, and Aggressiveness subscales range from 0 to 100, where higher score indicates worse severity than the average child with autism.
  The Social Approach, Expressive, and Learning Memory subscales range from 0 to 100, where higher score indicates better skills relative to the average child with autism.
  Scores reported in subscales. Scores were not reported as full scale.
Time Frame: Week 4 of Phase 1
Population: Data provided for participants who completed week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IGF-1, Week 4, Phase 1: Dose titration will be initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Doses may be decreased according to tolerability by 0.04 mg/kg per dose. Medication will be administered twice daily with meals, and pre-prandial glucose monitoring will be performed by parents at treatment initiation, prior to each injection, and until a well-tolerated dose is established.
- Placebo, Week 4, Phase 1: Placebo
  Placebo/saline: Placebo
Arm/Group | IGF-1, Week 4, Phase 1 | Placebo, Week 4, Phase 1
Number analyzed (Participants) | 1 | 2
score on a scale
  Sensory | 21 (NA) — N=1 therefore there is no measure of dispersion | 16 (14.1)
  Ritual | 9 (NA) — N=1 therefore there is no measure of dispersion | 13 (14.1)
  Social Pragmatic | 20 (NA) — N=1 therefore there is no measure of dispersion | 14 (0)
  Semantic Pragmatic | 19 (NA) — N=1 therefore there is no measure of dispersion | 0.5 (0.7)
  Arouse | 23 (NA) — N=1 therefore there is no measure of dispersion | 20.5 (6.4)
  Specific Fears | 13 (NA) — N=1 therefore there is no measure of dispersion | 25 (1.4)
  Aggressiveness | 7 (NA) — N=1 therefore there is no measure of dispersion | 30 (25.5)
  Social Approach | 75 (NA) — N=1 therefore there is no measure of dispersion | 31 (15.6)
  Expressive | 36 (NA) — N=1 therefore there is no measure of dispersion | 18.5 (20.5)
  Learning Memory | 0 (NA) — N=1 therefore there is no measure of dispersion | 8.5 (2.1)

3. Secondary Outcome: Social Pervasive Developmental Disorder-Behavior Inventory (PDDBI)
Description: as for outcome 2
Time Frame: Week 12 of Phase 1
Population: Data provided for participants who completed week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IGF-1: Dose titration will be initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Doses may be decreased according to tolerability by 0.04 mg/kg per dose. Medication will be administered twice daily with meals, and pre-prandial glucose monitoring will be performed by parents at treatment initiation, prior to each injection, and until a well-tolerated dose is established.
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 0 | 1
score on a scale
  Sensory |  | 9 (NA) — N=1 therefore there is no measure of dispersion
  Ritual |  | 4 (NA) — N=1 therefore there is no measure of dispersion
  Social Pragmatic |  | 16 (NA) — N=1 therefore there is no measure of dispersion
  Semantic Pragmatic |  | 8 (NA) — N=1 therefore there is no measure of dispersion
  Arouse |  | 12 (NA) — N=1 therefore there is no measure of dispersion
  Specific Fears |  | 22 (NA) — N=1 therefore there is no measure of dispersion
  Aggressiveness |  | 18 (NA) — N=1 therefore there is no measure of dispersion
  Social Approach |  | 59 (NA) — N=1 therefore there is no measure of dispersion
  Expressive |  | 27 (NA) — N=1 therefore there is no measure of dispersion
  Learning Memory |  | 15 (NA) — N=1 therefore there is no measure of dispersion

4. Secondary Outcome: Social Pervasive Developmental Disorder-Behavior Inventory (PDDBI)
Description: as for outcome 2
Time Frame: Week 4 of Phase 2
Population: Data provided for participants who completed week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale
  Sensory | 11 (NA) — N=1 therefore there is no measure of dispersion |
  Ritual | 2 (NA) — N=1 therefore there is no measure of dispersion |
  Social Pragmatic | 13 (NA) — N=1 therefore there is no measure of dispersion |
  Semantic Pragmatic | 5 (NA) — N=1 therefore there is no measure of dispersion |
  Arouse | 16 (NA) — N=1 therefore there is no measure of dispersion |
  Specific Fears | 10 (NA) — N=1 therefore there is no measure of dispersion |
  Aggressiveness | 10 (NA) — N=1 therefore there is no measure of dispersion |
  Social Approach | 52 (NA) — N=1 therefore there is no measure of dispersion |
  Expressive | 36 (NA) — N=1 therefore there is no measure of dispersion |
  Learning Memory | 14 (NA) — N=1 therefore there is no measure of dispersion |

5. Secondary Outcome: Social Pervasive Developmental Disorder-Behavior Inventory (PDDBI)
Description: as for outcome 2
Time Frame: Week 8 of Phase 2
Population: Data provided for participants who completed week 8. Data not provided by participant for one subscale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale
  Sensory | 5 (NA) — N=1 therefore there is no measure of dispersion |
  Ritual | 1 (NA) — N=1 therefore there is no measure of dispersion |
  Social Pragmatic: number analyzed (Participants) | 0 | 0
  Semantic Pragmatic | 9 (NA) — N=1 therefore there is no measure of dispersion |
  Arouse | 10 (NA) — N=1 therefore there is no measure of dispersion |
  Specific Fears | 7 (NA) — N=1 therefore there is no measure of dispersion |
  Aggressiveness | 6 (NA) — N=1 therefore there is no measure of dispersion |
  Social Approach | 60 (NA) — N=1 therefore there is no measure of dispersion |
  Expressive | 43 (NA) — N=1 therefore there is no measure of dispersion |
  Learning Memory | 14 (NA) — N=1 therefore there is no measure of dispersion |

6. Secondary Outcome: Repetitive Behavior
Description: Repetitive Behavior: Repetitive Behavior Scale (RBS) - Includes 43 items scored 0 (behavior does not occur), 1 (behavior occurs and is a mild problem), 2 (behavior occurs and is a moderate problem), 3 (behavior occurs and is a severe problem). Full scale from 0-129, with higher scores indicating worse outcomes.
Time Frame: Phase 1 - Week 4 and 12, Phase 2 - Week 4 and 8
Population: Data provided for participants who were on study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale
  Week 4 of Phase 1 | 31 (NA) — N=1 therefore there is no measure of dispersion | 44 (41.0)
  Week 12 of Phase 1: number analyzed (Participants) | 0 | 1
  Week 12 of Phase 1 |  | 11 (NA) — N=1 therefore there is no measure of dispersion
  Week 4 of Phase 2: number analyzed (Participants) | 1 | 0
  Week 4 of Phase 2 | 11 (NA) — N=1 therefore there is no measure of dispersion |
  Week 8 of Phase 2: number analyzed (Participants) | 1 | 0
  Week 8 of Phase 2 | 8 (NA) — N=1 therefore there is no measure of dispersion |

7. Secondary Outcome: Caregiver Strain
Description: Caregiver Strain Index - 21 question tool, with response 1 (not al all) - 5 (very much). Total score on scale from 21-105. Higher score indicates poorer health outcomes.
Time Frame: Phase 1 - Week 4 and 12, Phase 2 - Week 4 and 8
Population: Data provided for participants who were on study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale
  Week 4, Phase 1 | 71 (NA) — N=1 therefore there is no measure of dispersion | 87 (9.9)
  Week 12, Phase 1: number analyzed (Participants) | 0 | 1
  Week 12, Phase 1 |  | 73 (NA) — N=1 therefore there is no measure of dispersion
  Week 4, Phase 2: number analyzed (Participants) | 1 | 0
  Week 4, Phase 2 | 54 (NA) — N=1 therefore there is no measure of dispersion |
  Week 8, Phase 2: number analyzed (Participants) | 1 | 0
  Week 8, Phase 2 | 54 (NA) — N=1 therefore there is no measure of dispersion |

8. Secondary Outcome: Children's Yale-Brown Obsessive Compulsive Disorder Scale for Pervasive Developmental Disorders
Description: Clinician-rated interview designed to evaluate repetitive behavior in children with pervasive developmental disorders (PDDs). It is a modification of the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS), developed to assess typically-developing children with obsessive compulsive behavior. Because of language limitations in children with PDDs the CY-BOCS-PDD only includes the five compulsion items: Time Spent, Interference, Distress, Resistance of repetitive behavior, and Control of repetitive behavior. Each item is rated from 0 (none) through 4 (extreme), and scores can range from 0 to 20, with higher scores reflecting more severe symptoms. Usually a score 8 is considered clinically significant.
Time Frame: Phase 1 - Week 4 and 12, Phase 2 - Week 4 and 8
Population: data not collected
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: The Clinical Global Impression - Severity Scale (CGI-S)
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating. Full scale is 1 (normal, not at all ill) to 7 (extremely ill).
Time Frame: Phase 1 - Week 4 and 12, Phase 2 - Week 4 and 8
Population: Data provided for participants who were on study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale
  Week 4, Phase 1 | 5 (NA) — N=1 so no measure of dispersion | 5 (1.4)
  Week 12, Phase 1: number analyzed (Participants) | 0 | 1
  Week 12, Phase 1 |  | 4 (NA) — N=1 so no measure of dispersion
  Week 4, Phase 2: number analyzed (Participants) | 0 | 1
  Week 4, Phase 2 |  | 4 (NA) — N=1 so no measure of dispersion
  Week 8, Phase 2: number analyzed (Participants) | 1 | 0
  Week 8, Phase 2 | 4 (NA) — N=1 so no measure of dispersion |

10. Secondary Outcome: Vineland Adaptive Behavior Composite Score
Description: The Vineland Adaptive Behavior Scales, Second Edition (Survey Interview Form) yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning.
Time Frame: Baseline and Phase 1 Week 12
Population: Data collected at baseline and Week 12 and only for participants on study.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 1 | 2
T-score
  Baseline | 55 (NA) — N=1 therefore there is no measure of dispersion | 51 (8.5)
  Week 12, Phase 1: number analyzed (Participants) | 0 | 1
  Week 12, Phase 1 |  | 57 (NA) — N=1 therefore there is no measure of dispersion

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | IGF-1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGF-1 (N=2) | Placebo (N=2)
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Sleep disturbance (General disorders) | 2 | 1
Irritability (Psychiatric disorders) | 1 | 2
Bruising easily (Blood and lymphatic system disorders) | 0 | 1
Increased energy (General disorders) | 1 | 1
Aggression towards others (Psychiatric disorders) | 0 | 2
oppositional behavior (Psychiatric disorders) | 0 | 1
Eye blinking (Eye disorders) | 0 | 1
Canker sore (General disorders) | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0
Vomiting/diarrhea (Gastrointestinal disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Congestion/allergies (General disorders) | 2 | 0
Fever/congestion (General disorders) | 2 | 0
Tic- head shake (Psychiatric disorders) | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01970345/Prot_SAP_000.pdf